CLINICAL TRIAL: NCT06896682
Title: Cortisol and Obesity - A Vicious Cycle? Hypoglycemia After Bariatric Surgery - Association With Cortisol Metabolism?
Status: Not yet recruiting | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Charlotte Røn Stolberg, MD, PhD, Principal Investigator, Senior Registrar in Endocrinology, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: VEK Projekt-ID S-20250006
Record Dates: First submitted 2025-03-03; First posted 2025-03-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Postbariatric Hypoglycemia
Keywords: cortisol; bariatric surgery; postbariatric hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about how bariatric surgery affects the metabolism of cortisol.

The main question it aims to answer is whether changes in cortisol contribute to the development of reactive hypoglycemia?

100 individuals who have previously undergone bariatric surgery, are planned to be included.

DETAILED DESCRIPTION:
Purpose The project investigates how bariatric surgery affects the metabolism of cortisol. Additionally, it examines whether changes in cortisol contribute to the development of reactive hypoglycemia, a serious complication observed after bariatric surgery.

Study Visits

Visit 1:

At the first visit, participants sign an informed consent form, complete a medical history questionnaire, undergo measurements (height, weight), and have blood samples taken. They also undergo an adrenal stimulation test (ACTH test), receive a continuous glucose monitor (CGM), and complete a questionnaire about hypoglycemia symptoms.

The CGM is a small device that continuously measures blood glucose levels via a tiny sensor placed on the skin, typically on the arm or abdomen.

The ACTH test is performed after the participant has rested for at least 15 minutes. A synthetic hormone (Synacthen) is injected to stimulate the adrenal glands to produce cortisol. Blood samples are collected immediately before the injection and again 30 minutes afterward. The visit is expected to last approximately 1 hour.

Participants wear the CGM until the second visit and are instructed to collect 24-hour urine samples. If they experience hypoglycemia symptoms between visits, they take a saliva sample for cortisol measurement 5 minutes after symptom onset and another exactly 24 hours later.

Visit 2:

Ten days after the first visit, participants return for the second visit, where they submit their 24-hour urine and saliva samples. They then undergo a three-hour extended meal test.

This test consists of consuming a standardized liquid meal (200 ml Nutridrink, containing per 100 ml: 150 kcal, 5.8 g fat, 18.4 g carbohydrates, and 5.9 g protein). While undergoing the meal test, participants continue wearing the CGM, have blood samples taken at 30-minute intervals, and complete another questionnaire on hypoglycemia. This visit is expected to last 4 hours, bringing the total expected study time to 5 hours.

Monitoring and Reporting To ensure participant safety throughout the study, the following procedures will be implemented to manage potential complications.

Participants will be closely monitored during all procedures, including blood sampling, the ACTH test, and the meal test. Any side effects or complications will be documented and reported to the principal investigator.

Emergency Preparedness Emergency medical equipment, allergy management supplies, and trained nurses will be available during all visits. The nurses are trained to handle cases of post-bariatric hypoglycemia. In the event of severe allergic reactions or other acute complications, immediate medical treatment will be provided, and the principal investigator will be contacted immediately.

Informed Consent Participants will receive detailed information about potential risks and side effects before the study begins. They will be encouraged to report any discomfort or side effects immediately.

Follow-up Participants will have the opportunity to contact the principal investigator between and after visits if they experience any issues or have questions.

Protocol for Study Discontinuation If a participant experiences severe complications, their participation in the study will be discontinued, and they will receive appropriate medical care as outlined above, along with follow-up observation until they are in stable condition. The principal investigator will assess the situation and adjust the study protocol if necessary to prevent further complications.

Financial Aspects The project is funded through research grants from the Region of Southern Denmark. No financial compensation is provided to participants, except for reimbursement of transportation costs.

ELIGIBILITY:
Inclusion Criteria:

Participants must have undergone one of the following bariatric procedures at least 12 months prior:

* Roux-en-Y gastric bypass
* Gastric sleeve

Exclusion Criteria

* Pregnancy and breastfeeding
* Nephrotic syndrome (kidney disease with protein loss in urine), liver cirrhosis, or severe malnutrition, as these conditions reduce cortisol-binding globulin (CBG) levels, affecting total cortisol concentration
* Use of corticosteroid medications, such as prednisolone
* Use of opiod-containing medication
* Use of medications containing estrogen, such as hormone therapy for menopause
* Known adrenal disease affecting cortisol metabolism, including autonomous cortisol production and Cushing's syndrome
* Diabetes that does not require medical treatment
* Previously diagnosed reactive hypoglycemia after bariatric surgery requiring medical treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: postbariatric patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in serum cortisol during mixed meal test | 0, 30, 60, 90, 120, 150, 180 minutes (visit 2)
  cortisol at nadir glucose during the mixed meal test - cortisol at the start of the meal test

SECONDARY OUTCOMES:
ACTH test: Test of adrenal function | 0, 30 minutes
  0 min: Cortisol and corticotropin 30 min: Cortisol, corticotropin Δ Cortisol (30-minute cortisol - 0-minute cortisol) Bloodsamples
Cortisol hormone profile | 1 hour
  Bloodsamples of CBG, Cortisol, Cortisone
urinary cortisol: Ratio of cortisol/cortisone | 24 hour
  24-hour urinary cortisol: Ratio of cortisol/cortisone Urine sampling for 24 hour